CLINICAL TRIAL: NCT02277821
Title: Evaluation of the Action of the Stendo Pulsating Suit on Peripheral Microcirculation and on Central Blood Pressure in Essential Hypertension Patients Treated But Not Stabilized
Brief Title: Evaluation of Stendo Pulsating Suit on Microcirculation and Central Blood Pressure in Essential Hypertension Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stendo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-A00804-43
Record Dates: First submitted 2014-10-08; First posted 2014-10-29 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2014-10

CONDITIONS: Essential Hypertension
Keywords: Essential Hypertension; Central Blood Pressure; Microcirculation; Endothelium Stimulation
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stendo pulsating suit System (Experimental): One 20 minutes Stendo pulsating suit session will be applied to the patient.
  Interventions: Device: Stendo pulsating suit System

INTERVENTIONS:
Device: Stendo pulsating suit System — The Stendo system, a multilayer pulsatile inflatable suit is applied to the lower limbs and the abdomen. This device induces a sequential compartmentalized compression synchronized with each diastolic phase of the cardiac cycle, each phase evolving centripetally (lower limbs to abdomen).

SUMMARY:
The action of one Stendo pulsating suit session will be evaluated on 24 patients referred to the hypertension consultations for essential hypertension treated but not stabilized. The effect of one Stendo pulsating suit session system will be mainly assessed on the peripheral cutaneous microcirculation and on the central arterial pressure.

DETAILED DESCRIPTION:
The role of the endothelium in micro-vascular system is mediated by synthesis and release of numerous substances that act on the smooth muscle fibres. The release of these products is modulated, in turn, by various circulating molecules, by the autonomic nervous system and by local mechanical factors such as shear stress.

The essential hypertension is associated to increased risks of cardiovascular and stroke morbidity and mortality and constitutes a major cause of severe kidney failure. The essential hypertension is a complex and multi-factorial disease; the dysfunction of the endothelium is of a great importance in the physiopathology of this disease, concerning both the consequences of the increase of the blood pressure and the possible cause of the hypertension development.

The Stendo pulsating suit is expected to increase the cutaneous microcirculation measured by laser Doppler laser flowmetry and potentially to decrease the central blood pressure. Each patient will be his own witness and the clinical records will be assessed before, during when relevant, and after a pulsating suit session.

ELIGIBILITY:
Inclusion Criteria:

* Patient referred to the Hypertension Hospital Consultation for essential hypertension treated but not stabilized
* Patient with essential hypertension defined by a brachial arterial pressure of 140 ≤ Systolic Arterial Pressure < 180 mm Hg and/or 90 ≤ Diastolic Arterial - Pressure < 110 mm Hg
* Essential Hypertension confirmed by an ambulatory measure of the arterial pressure during 24 hours before the pre-inclusion visit
* Patients aged more than 40 and less than 70

Exclusion Criteria:

* Patient with secondary hypertension
* Patient with diabetes
* Patient with complete arrhythmia with atrial fibrillation
* Patient with an advanced obstructive arterial disease
* Patient with a recent and progressive deep venous thrombosis

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Peripheral microcirculation measured using Laser Doppler flowmetry | 35 minutes after the end of the Stendo session at D1 + 7 jours +/- 3
  Change in % of the peripheral cutaneous microcirculation using laser Doppler flowmetry after one Stendo pulsating suit session

SECONDARY OUTCOMES:
Humeral arterial pressure | 20 minutes after the end of Stendo session at D1 + 7 jours +/- 3
  Humeral arterial pressure using automatic measures with Dinamap device
Central blood pressure | Just after the end of the Stendo session.at D1 + 7 jours +/- 3
  Central blood pressure measured by applanation using an applanation tonometry device; Central pulse pressure, Augmentation Index and subendocardial viability ratio will also be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Guy AMAH, MD, Principal Investigator — Service de Physiologie Clinique - Explorations Fonctionnelles
Locations (1):
- Hôpital Lariboisière - Service de Physiologie Clinique - Explorations Fonctionnelles, Paris, France